CLINICAL TRIAL: NCT05096780
Title: Characterizing the Pharmacokinetic Profile of a Novel Encapsulated Caffeine Beverage and Associated Mood and Physiological Effects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEP-2110
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Alertness
Keywords: caffeine; beverage; energy; mood; encapsulated; Caffeine Research VAS

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Beverage 1 (Active Comparator): Free caffeine 160 mg
  Interventions: Other: Flavored caffeinated beverage
- Beverage 2 (Experimental): Encapsulated caffeine 160 mg
  Interventions: Other: Flavored caffeinated beverage
- Beverage 3 (Active Comparator): Free caffeine 250 mg
  Interventions: Other: Flavored caffeinated beverage
- Beverage 4 (Experimental): Encapsulated caffeine 250 mg
  Interventions: Other: Flavored caffeinated beverage

INTERVENTIONS:
Other: Flavored caffeinated beverage — 16.9 oz (500 cc), carbonated, zero calorie

SUMMARY:
This study is designed to compare self-reported mood states for encapsulated caffeine compared to dose-matched free caffeine, when consumed as a ready-to-drink beverage in healthy subjects. Additionally, this study will characterize the plasma caffeine pharmacokinetic profile for the encapsulated and free caffeine beverages. Two different caffeine levels, 160 and 250 mg will be included, which represent more common caffeine consumption from typical energy drinks.

The primary outcomes are alertness ratings from the Caffeine Research visual analog scale (VAS) and PK parameters over 12 hours. Secondary outcomes are Caffeine Research VAS scores (beyond alertness), three other symptom VAS scores, and vital signs for safety.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male and female volunteers aged 18 to 55 years
2. Have a BMI of 18 to 32.49 kg/m2 (inclusive)
3. Are regular caffeine consumers (average 1 to 3 caffeine-containing beverages per day, not to exceed 400 mg/ per day)
4. Willing to commit to 4 long test days (~15-16 hrs)
5. Able to comprehend and willing to sign an Informed Consent Form (ICF)
6. Willing to avoid caffeine-containing products for ≥48 hrs prior to visits and until the completion of each test visit
7. Willing to avoid alcohol for ≥24 hrs prior to visits
8. Willing to fast 10 hrs prior to visits
9. Willing to stick to their usual dietary patterns and avoid grapefruit
10. Willing to stick to their usual physical activity level throughout the study
11. Willing to stick to their usual sleep pattern
12. No participation in any clinical trial within the past 30 days and throughout this study, or any PEP protocol within the past 6 months

Exclusion Criteria:

Subjects will be excluded from the study if they have:

1. Reported history or clinical manifestations of significant metabolic (including type1 or type 2 diabetes mellitus), hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, urological, neurological, or psychiatric disorders unless deemed clinically not significant by investigator
2. Current or recent history (<30 days prior to Screening) of a clinically significant bacterial, fungal, or mycobacterial infection
3. Current clinically significant viral infection
4. History of malignancy, with the exception of cured basal cell or squamous cell carcinoma of the skin
5. Are pregnant or breastfeeding or planning to become pregnant
6. Resting heart rate less than 45 bpm or greater than 100 bpm
7. History of unstable ischemic heart disease or uncontrolled hypertension (blood pressure greater than or equal to 50/90 mm Hg)
8. History of significant surgery that may affect absorption of caffeine. Appendectomy and/or cholecystectomy will be allowed
9. Presence of a malabsorption syndrome possibly affecting drug/Product absorption (e.g., Crohn's disease or chronic pancreatitis)
10. Extreme dietary habits, including but not limited to intentional consumption of a high fiber diet, gluten-free, low-carb, vegan, ketogenic
11. History of alcoholism or drug addiction within 1 year prior to Screening, or current alcohol or drug use that, in the opinion of the investigator, will interfere with the subject's ability to comply with the dosing schedule and study evaluations
12. One or more tobacco-containing or nicotine-containing product occasions per month on average, or use of such products within 48 hours prior to dosing of each study period
13. Use of any prescription or nonprescription drugs (including vitamins, minerals, and phytotherapeutic, herbal, or plant-derived preparations) is prohibited within 7 days prior to the dose of study product, unless deemed acceptable by the Investigator
14. Use of any medication known to have an interaction with caffeine including oral contraceptives (e.g., medications metabolized via the CYP1A2 pathway)
15. Donation of blood in excess of 500 ml within 4 weeks prior to study entry or of plasma within 2 weeks prior to Screening
16. Receipt of blood products within 3 months prior to study entry
17. Subjects who, in the opinion of the investigator, are unable or unlikely to comply with the dosing schedule and study evaluations

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-02-06 (Actual); Study Completion 2022-02-06 (Actual)

PRIMARY OUTCOMES:
Alertness | Changes from pre-dose baseline to 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours post beverage ingestion
  A self-reported mood measurement from the Caffeine Research Visual Analog Scale (VAS) rated from 0 (not at all) to 100 mm (extremely alert), to compare dose-matched free caffeine to encapsulated caffeine. Longer-lasting alertness would be a benefit.
Plasma caffeine PK profile of (AUC0-t, AUC0-inf) | Changes from pre-dose baseline to 12 hours after the first sip of beverage.
  Plasma sampling at 19 time points: Pre-dose baseline, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 9, 10, 11 and 12 hours post first sip of beverage ingestion to characterize dose-matched free caffeine compared to encapsulated caffeine for plasma caffeine (AUC0-t, AUC0-inf)
Plasma caffeine PK profile of peak caffeine concentration (Cmax) | Changes from pre-dose baseline to 12 hours after the first sip of beverage.
  Plasma sampling at 19 time points: Pre-dose baseline, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 9, 10, 11 and 12 hours post first sip of beverage ingestion to characterize dose-matched free caffeine compared to encapsulated caffeine for plasma caffeine peak caffeine concentration (Cmax)
Plasma caffeine PK profile of time to maximal plasma caffeine concentration (Tmax) | Changes from pre-dose baseline to 12 hours after the first sip of beverage.
  Plasma sampling at 19 time points: Pre-dose baseline, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 9, 10, 11 and 12 hours post first sip of beverage ingestion to characterize dose-matched free caffeine compared to encapsulated caffeine for plasma caffeine time to maximal plasma caffeine concentration (Tmax)
Plasma caffeine PK profile of half-life (t1/2) | Changes from pre-dose baseline to 12 hours after the first sip of beverage.
  Plasma sampling at 19 time points: Pre-dose baseline, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 9, 10, 11 and 12 hours post first sip of beverage ingestion to characterize dose-matched free caffeine compared to encapsulated caffeine for plasma caffeine half-life (t1/2)
Plasma caffeine PK profile of plasma caffeine concentration by time | Changes from pre-dose baseline to 12 hours after the first sip of beverage.
  Plasma sampling at 19 time points: Pre-dose baseline, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 9, 10, 11 and 12 hours post first sip of beverage ingestion to characterize dose-matched free caffeine compared to encapsulated caffeine for plasma caffeine concentration by time

SECONDARY OUTCOMES:
The 6 other Caffeine Research Visual Analog Scale (VAS) symptom ratings besides alertness | Changes from pre-dose baseline to 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours post beverage ingestion
  Self-reported Caffeine Research Visual Analog Scale (VAS) ratings from 0-100 mm representing the full range of each dimension (relaxed, jittery, tired, tense, headache, overall mood) to compare dose-matched free caffeine to encapsulated caffeine. More relaxed, less jittery, less tired, less tense, no headache and better mood would be better.
3 additional other symptoms Visual Analog Scale (VAS) ratings | Changes from pre-dose baseline to 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours post beverage ingestion
  Self-reported caffeine symptoms (lightheaded, irritable, pounding heartbeat) rated on a Visual Analog Scale (VAS) from 0 (not at all) to 100 mm (extremely) to compare dose-matched free caffeine to encapsulated caffeine. Absence of these would be better.
Blood pressure | Changes from pre-dose baseline to 2 and 6 hours post beverage ingestion
  Vital sign for safety monitoring. Resting blood pressures within normal limits would be better.
Heart rate | Changes from pre-dose baseline to 2 and 6 hours post beverage ingestion
  Vital sign for safety monitoring. Resting heart rates within normal limits would be better.

CONTACTS AND LOCATIONS:
Overall Officials: Swarna Yadlapalli, MD, Principal Investigator — Medical Director, Axis Clinicals
Locations (1):
- AXIS Clinicals, Dilworth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No